CLINICAL TRIAL: NCT01593696
Title: Phase I Study of T Cells Expressing an Anti-CD19 Chimeric Receptor in Children and Young Adults With B Cell Malignancies
Brief Title: Anti-CD19 White Blood Cells for Children and Young Adults With B Cell Leukemia or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nirali N. Shah, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 120112; 12-C-0112
Record Dates: First submitted 2012-05-05; First posted 2012-05-08 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: ALL; B Cell Lymphoma; Leukemia; Large Cell Lymphoma; Non-Hodgkin Lymphoma
Keywords: CD 19 Expressing B Cells; B Cell Lymphoma; ALL; Anti-CD19 Chimeric Antigen Receptor; Adoptive Immunotherapy
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lymphodepleting regimen of Fludarabine and Cyclophosphamide (Experimental): Lymphodepleting regimen of Fludarabine and Cyclophosphamide.
  Interventions: Biological: Anti-Cluster of Differentiation (CD)19-Chimeric antigen receptor (CAR)
- Intensive standard of care chemotherapy (Experimental): Intensive standard of care chemotherapy, in lieu of the lymphodepleting chemotherapy regimen, to decrease tumor burden in preparation for the administration of the Chimeric antigen receptor (CAR) T cells.
  Interventions: Biological: Anti-Cluster of Differentiation (CD)19-Chimeric antigen receptor (CAR)

INTERVENTIONS:
Biological: Anti-Cluster of Differentiation (CD)19-Chimeric antigen receptor (CAR) — Cells extracted, followed by induction chemotherapy before Cluster of Differentiation (CD)19-Chimeric antigen receptor (CAR) infusion (dose escalation.)

SUMMARY:
Background:

- Although progress has been made in treating children with B-cell cancers such as leukemia or lymphoma, many children do not respond to the standard treatments. One possible treatment involves collecting white blood cells called T cells from the person with cancer and modifying the cells to attack the B-cell cancer. The cells can then be given back to the participant. This study will use T cells that have been modified to attack the cluster of differentiation 19 (CD19) protein, which is found on the surface of some B-cell cancers.

Objectives:

- To see if anti-CD19 modified white blood cells are a safe and effective treatment for children and young adults with advanced B-cell cancer.

Eligibility:

* Children and young adults between 1 and 30 years of age who have B-cell cancer (leukemia or lymphoma) that has not responded to standard treatments.
* The leukemia or the lymphoma must have the CD19 protein.
* There must be adequate organ function.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies or bone marrow biopsies may be performed depending on the type of cancer.
* Participants will undergo a process where white blood cells are collected, called apheresis. These cells will be modified to contain the anti-CD19 gene.
* Participants will have 3 days of chemotherapy to prepare their immune system to accept the modified cells.
* Participants will receive an infusion of their own modified white blood cells. They will remain in the hospital until they have recovered from the treatment.
* Participants will have frequent follow-up visits to monitor the outcome of the treatment.
* If the participant benefits from the treatment, then he/she may have the option for another round of treatment.

DETAILED DESCRIPTION:
Background:

Chimeric antigen receptors (CAR) that recognize the cluster of differentiation 19(CD19) antigen have been constructed and are in clinical trials at several institutions. In this trial, the Pediatric Oncology Branch (POB) will utilize a chimeric receptor containing the signaling domains of cluster of differentiation 28 (CD28) and cluster of differentiation 3 (CD3)-zeta, currently under study in the Center for Cancer Research (CCR) in adults, for children and young adults with CD19 expressing malignancies.

In co-cultures with CD19-expressing acute lymphoblastic leukemia cells, anti-CD19-CAR-transduced T cells show robust killing, and in xenograft models, can rapidly clear CD19- expressing ALL cell lines.

Objectives:

1. Primary: To determine the safety and feasibility of administering escalating doses of anti-CD19-CAR engineered peripheral blood lymphocytes in two strata (prior allogeneic stem cell transplant [SCT] vs. no prior SCT) of children and young adults with B cell malignancies following a cyclophosphamide/fludarabine preparative regimen. COMPLETED March 2014.
2. Primary: To determine the safety of administering cells in two groups of children and young adults with B-cell malignancies expressing CD19:

   * Arm 1 - Patients without high-burden disease or patients for whom chemotherapy toxicity is a concern will receive standard preparative regimen.
   * Arm 2 - Patients with high-burden disease who receive standard chemotherapy to reduce burden, (defined as patients with ALL who have M3 bone marrow blasts and/or presence of peripheral blood blasts on routine complete blood count (CBC), or patients with lymphoma).
3. Primary: To determine the feasibility of administering anti-CD19 CAR transduced T cells within 21 days of the target date in children and young adults with B-cell malignancies expressing CD19 enrolled on arm 2: Patients with high-burden disease who receive standard chemotherapy to reduce burden.

1) Secondary: 1) To determine if the administration of anti-CD19-CAR engineered peripheral blood lymphocytes can mediate antitumor effects in children with B cell high-burden disease after standard chemotherapy, or in patients without high-burden disease who receive standard preparative regimen. 2) To evaluate the ability of CRS treatment algorithm to reduce the incidence of Grade 4 Cytokine Release Syndrome (CRS) to less than or equal to 10% of patients. 3) To measure persistence of adoptively-transferred anti-CD19-CAR-transduced T cells in the blood, bone marrow and cerebrospinal fluid (CSF) of patients. 4) To describe the toxicity of administration of anti-CD19-CAR engineered peripheral blood lymphocytes in children and young adults with central nervous system (CNS) disease.

Eligibility:

Patients 1-30 years of age, at least 15 kg, with a CD19-expressing B-cell malignancy that has recurred after or not responded to one or more standard chemotherapy-containing regimens for their malignancy and is deemed incurable by standard therapy. Patients with a history of allogeneic stem cell transplant who meet all eligibility criteria are eligible to participate.

Design:

* PBMC will be obtained by leukapheresis. Anti-CD19 CAR T cells will be manufactured from fresh or frozen peripheral blood mononuclear cells (PBMCs). On Day -7, PBMC will be enriched for cluster of differentiation 3 (CD3)+ cells and cultured in the presence of anti-CD3/-cluster of differentiation 28 (CD28) beads followed by retroviral vector supernatant containing the anti-cluster of differentiation 19 (CD19) CAR. Total culture time is approximately 7-14 days.
* Patients will be divided into the 2 groups listed above.

Arm 1: Patients will begin preparative regimen comprising fludarabine 25 mg/m(2) on Days -4, -3 and -2 and cyclophosphamide 900 mg/m(2) on day -2.

Arm 2: Patients with high-disease burden will be treated with intensive standard of care chemotherapy to decrease disease burden during cell manufacturing.

* All patients: The CD19-CAR cells will be infused on Day 0, with up to a 72h delay allowed for fresh cells or a 21 day delay if cells are cryopreserved, if needed for resolution of clinical toxicities or to generate adequate cell numbers.
* The previously determined maximum tolerated dose (MTD) of 1 X 10(6) will be administered intravenously.
* Patients will be monitored for toxicity, response and T cell persistence.

ELIGIBILITY:
* INCLUSION CRITERIA
* Patient must have a cluster of differentiation 19 (CD19)-expressing B cell ALL or lymphoma and must have relapsed or refractory disease after at least one standard chemotherapy and one salvage regimen. In view of the principal investigator (PI) and the primary oncologist, there must be no available alternative curative therapies and subjects must be either ineligible for allogeneic stem cell transplant (SCT), have refused SCT, or have disease activity that prohibits SCT at this time.
* CD19 expression must be detected on greater than 15% of the malignant cells by immunohistochemistry or greater than 30% by flow cytometry in a Clinical Laboratory Improvement Amendments (CLIA) approved test in the Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI), National Institutes of Health (NIH), or from the referring institution or reference laboratory. The choice of whether to use flow cytometry or immunohistochemistry will be determined by what is the most easily available tissue sample in each patient. In general immunohistochemistry will be used for lymph node biopsies, flow cytometry will be used for peripheral blood and bone marrow samples.
* Patients must have measurable or evaluable disease at the time of enrollment, which may include any evidence of disease including minimal residual disease detected by flow cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis.
* Greater than or equal to 1 year of age (and at least 15 kg) and less than or equal to 30 years of age.
* Adequate absolute CD3 count estimated to be required to obtain target cell dose based on discussion with Department of Transfusion Medicine (DTM) apheresis and Cell Processing Section, DTM.
* Subjects with the following central nervous system (CNS) status are eligible only in the absence of neurologic symptoms suggestive of CNS leukemia, such as cranial nerve palsy:

  * CNS 1, defined as absence of blasts in cerebral spinal fluid (CSF) on cytospin preparation, regardless of the number of WBCs;
  * CNS 2, defined as presence of < 5/uL white blood cells (WBCs) in CSF and cytospin positive for blasts, or > 5/uL WBCs but negative by Steinherz/Bleyer algorithm
  * CNS3 with marrow disease who has failed salvage systemic and intensive IT chemotherapy (and therefore not eligible for radiation)
  * Patients with isolated CNS relapse will be eligible if they have previously been treated with cranial radiation (at least centigray (cGy)).
* Ability to give informed consent. For subjects <18 years old their legal guardian must give informed consent. Pediatric subjects will be included in age appropriate discussion and verbal assent will be obtained for those greater than or equal to 12 years of age, when appropriate.
* Clinical performance status: Patients > 10 years of age: Karnofsky greater than or equal to 50%; Patients less than or equal to 10 years of age: Lansky scale greater than or equal to 50%. Subjects who are unable to walk because of paralysis, but who are upright in a wheelchair will be considered ambulatory for the purpose of calculating the performance score.
* Patients of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four months after receiving the preparative regimen.
* Females of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects on the fetus.
* Cardiac function: Left ventricular ejection fraction greater than or equal to 40% by multi-gated acquisition scan (MUGA) or cardiac magnetic resonance imaging (MRI), or fractional shortening greater than or equal to 28% by echocardiogram (ECHO) or left ventricular ejection fraction greater than or equal to 50% by ECHO.
* Patients with history of allogeneic stem cell transplantation are eligible if at least 100 days post-transplant, if there is no evidence of active graft versus host disease (GVHD) and no longer taking immunosuppressive agents for at least 30 days prior to enrollment.

EXCLUSION CRITERIA

Subjects meeting any of the following criteria are not eligible for participation in the study:

* Recurrent or refractory ALL limited to isolated testicular disease.
* Hepatic function: Inadequate liver function defined as total bilirubin > 2x upper limit of normal (ULN) (except in the case of subjects with documented Gilbert's disease > 3x ULN) or transaminase (alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 20x ULN based on age and laboratory specific normal ranges;
* Renal function: Greater than age-adjusted normal serum creatinine (see below) and a creatinine clearance < 60 mL/min/1.73 m^2.

  * Age:

    * <= 5 yrs (Maximum Serum Creatinine = 0.8 mg/dL)
    * 5 < age <=10 yrs (Maximum Serum Creatinine =1.0 mg/dL)
    * > 10 yrs (Maximum Serum Creatinine = 1.2 mg/dL)
* Hematologic function:

  * Absolute neutrophil count (ANC) < 750/microliter, or platelet count < 50,000/microliter, if these cytopenias are not judged by the investigator to be due to underlying disease (i.e. potentially reversible with anti-neoplastic therapy);
  * A subject will not be excluded because of pancytopenia greater than or equal to Grade 3 if it is due to disease, based on the results of bone marrow studies.
* Hyperleukocytosis (greater than or equal to 50,000 blasts/microliter) or rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy;
* Pregnant or breast-feeding females;
* Recent prior therapy:

  * Systemic chemotherapy less than or equal to 2 weeks (6 weeks for nitrosoureas) or radiation therapy less than or equal to 3 weeks prior to apheresis;

Exceptions:

* There is no time restriction in regard to prior intrathecal chemotherapy provided there is complete recovery from any acute toxic effects of such;
* Subjects receiving hydroxyurea may be enrolled provided there has been no increase in dose for at least 2 weeks prior to starting apheresis;
* Patients who relapse while receiving standard ALL maintenance chemotherapy will not be required to have a waiting period before entry onto this study provided they meet all other eligibility criteria;
* Subjects receiving steroid therapy at physiologic replacement doses only are allowed provided there has been no increase in dose for at least 2 weeks prior to starting apheresis;
* For radiation therapy: Radiation therapy must have been completed at least 3 weeks prior to enrollment, with the exception that there is no time restriction if the volume of bone marrow treated is less than 10% and also the subject has measurable/evaluable disease outside the radiation port.

  * Other anti-neoplastic investigational agents currently or within 30 days prior to apheresis (i.e. start of protocol therapy);
  * Subjects must have recovered from the acute side effects of their prior therapy, such that eligibility criteria are met. Cytopenias deemed to be disease-related and not therapy-related are exempt from this exclusion.

    * Human immunodeficiency virus/hepatitis B virus/Hepatitis C virus (HIV/HBV/HCV) Infection:
* Seropositive for HIV antibody. (Patients with HIV are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy in the future should study results indicate effectiveness.)
* Seropositive for hepatitis C or positive for Hepatitis B surface antigen (HbsAG).

  * Monoclonal antibody therapy administered within 30 days of the agent prior to apheresis;
  * Uncontrolled, symptomatic, intercurrent illness including but not limited to infection, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the principal investigator (PI) would pose an unacceptable risk to the subject;
  * Second malignancy other than in situ carcinoma of the cervix, unless the tumor was treated with curative intent at least two years previously and subject is in remission;
  * History of severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biologic composition to any agents used in study or in the manufacturing of the cells (i.e. gentamicin);

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2012-06-29 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2017-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirali N Shah, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kowolik CM, Topp MS, Gonzalez S, Pfeiffer T, Olivares S, Gonzalez N, Smith DD, Forman SJ, Jensen MC, Cooper LJ. CD28 costimulation provided through a CD19-specific chimeric antigen receptor enhances in vivo persistence and antitumor efficacy of adoptively transferred T cells. Cancer Res. 2006 Nov 15;66(22):10995-1004. doi: 10.1158/0008-5472.CAN-06-0160. PMID 17108138
- [Background] Kochenderfer JN, Wilson WH, Janik JE, Dudley ME, Stetler-Stevenson M, Feldman SA, Maric I, Raffeld M, Nathan DA, Lanier BJ, Morgan RA, Rosenberg SA. Eradication of B-lineage cells and regression of lymphoma in a patient treated with autologous T cells genetically engineered to recognize CD19. Blood. 2010 Nov 18;116(20):4099-102. doi: 10.1182/blood-2010-04-281931. Epub 2010 Jul 28. PMID 20668228
- [Background] Morgan RA, Yang JC, Kitano M, Dudley ME, Laurencot CM, Rosenberg SA. Case report of a serious adverse event following the administration of T cells transduced with a chimeric antigen receptor recognizing ERBB2. Mol Ther. 2010 Apr;18(4):843-51. doi: 10.1038/mt.2010.24. Epub 2010 Feb 23. PMID 20179677
- [Derived] Silbert SK, Madan S, Holland EM, Steinberg SM, Little L, Foley T, Epstein M, Sarkisian A, Lee DW, Nikitina E, Kakumanu S, Ruppin E, Shalabi H, Yates B, Shah NN. A comprehensive analysis of adverse events in the first 30 days of phase 1 pediatric CAR T-cell trials. Blood Adv. 2023 Sep 26;7(18):5566-5578. doi: 10.1182/bloodadvances.2023009789. PMID 37486616
- [Derived] Shalabi H, Martin S, Yates B, Wolters PL, Kaplan C, Smith H, Sesi CR, Jess J, Toledo-Tamula MA, Struemph K, Delbrook CP, Khan OI, Mackall CL, Lee DW, Shah NN. Neurotoxicity following CD19/CD28zeta CAR T-cells in children and young adults with B-cell malignancies. Neuro Oncol. 2022 Sep 1;24(9):1584-1597. doi: 10.1093/neuonc/noac034. PMID 35148417
- [Derived] Molina JC, Steinberg SM, Yates B, Lee DW, Little L, Mackall CL, Shalabi H, Shah NN. Factors Impacting Overall and Event-Free Survival following Post-Chimeric Antigen Receptor T Cell Consolidative Hematopoietic Stem Cell Transplantation. Transplant Cell Ther. 2022 Jan;28(1):31.e1-31.e9. doi: 10.1016/j.jtct.2021.10.011. Epub 2021 Oct 20. PMID 34687939
- [Derived] Shah NN, Lee DW, Yates B, Yuan CM, Shalabi H, Martin S, Wolters PL, Steinberg SM, Baker EH, Delbrook CP, Stetler-Stevenson M, Fry TJ, Stroncek DF, Mackall CL. Long-Term Follow-Up of CD19-CAR T-Cell Therapy in Children and Young Adults With B-ALL. J Clin Oncol. 2021 May 20;39(15):1650-1659. doi: 10.1200/JCO.20.02262. Epub 2021 Mar 25. PMID 33764809
- [Derived] Shalabi H, Sachdev V, Kulshreshtha A, Cohen JW, Yates B, Rosing DR, Sidenko S, Delbrook C, Mackall C, Wiley B, Lee DW, Shah NN. Impact of cytokine release syndrome on cardiac function following CD19 CAR-T cell therapy in children and young adults with hematological malignancies. J Immunother Cancer. 2020 Sep;8(2):e001159. doi: 10.1136/jitc-2020-001159. PMID 32883871
- [Derived] Lee DW, Kochenderfer JN, Stetler-Stevenson M, Cui YK, Delbrook C, Feldman SA, Fry TJ, Orentas R, Sabatino M, Shah NN, Steinberg SM, Stroncek D, Tschernia N, Yuan C, Zhang H, Zhang L, Rosenberg SA, Wayne AS, Mackall CL. T cells expressing CD19 chimeric antigen receptors for acute lymphoblastic leukaemia in children and young adults: a phase 1 dose-escalation trial. Lancet. 2015 Feb 7;385(9967):517-528. doi: 10.1016/S0140-6736(14)61403-3. Epub 2014 Oct 13. PMID 25319501
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0112.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%); Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%): Lymphodepleting regimen of Fludarabine and Cyclophosphamide.
  Anti-Cluster of Differentiation (CD)19-Chimeric antigen receptor (CAR): Cells extracted, followed by induction chemotherapy before CD19-CAR infusion.
  Follow-up through at least 28 days after CD19 CAR infusion.
- Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%); Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%): Intensive lymphodepleting chemotherapy, in lieu of the standard lymphodepleting chemotherapy regimen, to decrease tumor burden in preparation for the administration of the Chimeric antigen receptor (CAR) T cells.
  Anti-Cluster of Differentiation (CD)19- Chimeric antigen receptor (CAR): Cells extracted, followed by induction chemotherapy before CD19-CAR infusion.
  Follow-up through at least 28 days after CD19 CAR infusion.
Period: Dose Escalation
Arm/Group | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%)
Started | 16 | 5 | 0 | 0
Prior Transplant | 7 | 1 | 0 | 0
No Prior Transplant | 9 | 4 | 0 | 0
Completed | 14 | 5 | 0 | 0
Not Completed | 2 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%)
Started | 0 | 0 | 16 | 16
Completed | 0 | 0 | 15 | 16
Not Completed | 0 | 0 | 1 | 0
Not completed — Fungal infection | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%); Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%); Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%): Lymphodepleting regimen of Fludarabine and Cyclophosphamide. Anti-Cluster of Differentiation (CD)19-Chimeric antigen receptor (CAR): Cells extracted, followed by induction chemotherapy before CD19-CAR infusion.
- Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%): Intensive lymphodepleting chemotherapy, in lieu of the standard lymphodepleting chemotherapy regimen, to decrease tumor burden in preparation for the administration of the Chimeric antigen receptor (CAR) T cells.
  Anti-Cluster of Differentiation (CD)19- Chimeric antigen receptor (CAR): Cells extracted, followed by induction chemotherapy before CD19-CAR infusion.
- Total: Total of all reporting groups
Arm/Group | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Total
Number analyzed (Participants) | 16 | 5 | 16 | 16 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 4 | 14 | 10 | 38
  Between 18 and 65 years | 6 | 1 | 2 | 6 | 15
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.75 (6.3) | 12.7 (6.09) | 13.04 (4.98) | 15.06 (7.92) | 14.29 (6.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 2 | 3 | 12
  Male | 9 | 5 | 14 | 13 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 6 | 6 | 19
  Not Hispanic or Latino | 12 | 2 | 10 | 10 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 16 | 4 | 10 | 11 | 41
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 16 | 5 | 16 | 16 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Preparative Chemotherapy Followed by Cluster of Differentiation (CD)19-Chimeric Antigen Receptor (CAR): CD19 CAR T-cells With < Grade 4 Cytokine Release Syndrome
Description: Participants with B cell malignancies who received preparative chemotherapy followed by CD19 CAR T-cells with < Grade 4 cytokine release syndrome.
Time Frame: Beginning of preparative regimen through Day 28 after CD19 CAR infusion
Population: Only 15/16 subjects were analyzed in Phase 2, Arm 1 because one subject did not received CAR cell infusion and therefore could not be evaluated for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%)
Number analyzed (Participants) | 16 | 5 | 15 | 16
Participants | 14 | 4 | 14 | 15

2. Primary Outcome: Number of Participants in Which the Prescribed Dose of Cluster of Differentiation (CD)19-Chimeric Antigen Receptor (CAR): CD19 CAR T-cells Were Successfully Manufactured
Description: Participants who had T-cells collected by apheresis and subsequently had the amount of CAR T-cells manufactured as prescribed by the dose level they were enrolled in.
Time Frame: Apheresis through completion of CAR manufacturing process, approximately 2 weeks
Population: Per protocol, only patients treated in Phase 1 were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%)
Number analyzed (Participants) | 16 | 5 | 0 | 0
Participants | 15 | 4 | 0 | 0

3. Secondary Outcome: Number of Participants Who Were Administered Intensive Chemotherapy Prior to Cluster of Differentiation (CD)19-Chimeric Antigen Receptor (CAR): CD19 CAR Infusion
Description: Participants who were administered intensive chemotherapy prior to Cluster of Differentiation (CD)19-Chimeric antigen receptor (CAR): CD19 CAR infusion and received CAR cells within 21 days of the planned infusion date.
Time Frame: 21 days of target date
Population: Per protocol, only participants on Phase 2, Arm 2 were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%)
Number analyzed (Participants) | 0 | 0 | 0 | 16
Participants | 0 | 0 | 0 | 16

4. Secondary Outcome: Mean Percentage Cluster of Differentiation 19 (CD19) - Chimeric Antigen-Receptor (CAR) T-Cells in Blood, Bone Marrow (BM) and Cerebrospinal Fluid (CSF)
Description: Measure persistence of adoptively-transferred anti-CD19-CAR transduced T cells (defined by percent of CD19 CAR T-cells) in the blood and where possible the bone marrow and Cerebrospinal Fluid (CSF) of patients by flow cytometry assay.
Time Frame: 28 days (+/- 4 days) after infusion of CD19 CAR T-cells
Population: Ph 1, Arm 1: BM analyzed in 13/16 subjects & CSF in 14/16 subjects as results not available in additional subjects. Ph 2, Arm 1: 14/16 subjects analyzed as 1 not infused & 1 developed PD. One additional subject didn't have BM/CSF results. Ph 2, Arm 2: 14/16 subjects analyzed as 2 developed PD. Two additional patients didn't have BM/CSF results.
Measure: Mean (Standard Deviation); unit: Percentage T-cells
Arm/Group | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%)
Number analyzed (Participants) | 16 | 5 | 14 | 14
Percentage T-cells
  Peripheral blood | 0.279 (0.712) | 0.122 (0.239) | 0.343 (1.022) | 0.897 (1.871)
  Bone marrow: number analyzed (Participants) | 13 | 5 | 13 | 12
  Bone marrow | 0.459 (0.781) | 0.554 (0.979) | 0.552 (1.308) | 0.814 (1.775)
  Cerebrospinal fluid: number analyzed (Participants) | 14 | 5 | 13 | 12
  Cerebrospinal fluid | 3.186 (5.304) | 1.825 (2.943) | 7.192 (16.728) | 14.742 (16.301)

5. Secondary Outcome: Number of Patients With a Complete Response (CR)
Description: Complete Response (CR) was assessed by bone marrow evaluation was I defined as <5% leukemic blasts.
Time Frame: Day 28 (+/- 4 days) after CD19 CAR infusion
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%)
Number analyzed (Participants) | 16 | 5 | 15 | 16
Participants | 10 | 4 | 11 | 6

6. Secondary Outcome: Number of Participants With Grade 4 Cytokine Release Syndrome (CRS)
Description: Participants with Grade 4 Cytokine Release Syndrome (CRS). CRS is defined as a clinical syndrome that may occur after cell therapy due to the release of cytokines (substances secreted by immune cells) into the body's blood stream.
Time Frame: Day 28 (+/- 4 days) after CD19 CAR infusion.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%)
Number analyzed (Participants) | 16 | 5 | 15 | 16
Participants | 2 | 1 | 1 | 1

7. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, from 1.5 months up to 3.1 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%)
Number analyzed (Participants) | 16 | 5 | 16 | 16
Participants | 16 | 5 | 16 | 16

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, from 1.5 months up to 3.1 years.
Arm/Group | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%)
All-Cause Mortality (participants affected / at risk) | 10/16 | 3/5 | 5/16 | 11/16
Serious Adverse Events (participants affected / at risk) | 6/16 | 2/5 | 1/16 | 5/16
Other Adverse Events (participants affected / at risk) | 16/16 | 5/5 | 16/16 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) (N=16) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) (N=5) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) (N=16) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) (N=16)
Cytokine release syndrome (Immune system disorders) | 3 (3) | 1 (1) | 1 (1) | 4 (9)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, biventricular dilatation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, L deviated gaze (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, increased ventricle size (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, dilated cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, elevated RVSP (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, global systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, intraventricular hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, ventriculomegaly (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, paraplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) (N=16) | Phase 1, Arm 2 - 3 x 10E6 Transduced T Cells/kg (+/- 20%) (N=5) | Phase 2, Arm 1 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) (N=16) | Phase 2, Arm 2 - 1 x 10E6 Transduced T Cells/kg (+/- 20%) (N=16)
Acoustic nerve disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 6 (10) | 5 (10) | 12 (21) | 14 (67)
Acute kidney injury (Renal and urinary disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (7) | 2 (3)
Alanine aminotransferase increased (Investigations) | 6 (22) | 2 (2) | 11 (39) | 12 (30)
Alkaline phosphatase increased (Investigations) | 4 (13) | 2 (2) | 5 (12) | 7 (12)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 11 (47) | 4 (19) | 14 (61) | 14 (139)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 2 (2) | 5 (8)
Anxiety (Psychiatric disorders) | 2 (3) | 0 (0) | 3 (5) | 7 (10)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 8 (32) | 2 (3) | 9 (48) | 14 (45)
Blood and lymphatic system disorders - Other, Total CO2 low (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (5)
Blood bilirubin increased (Investigations) | 4 (10) | 2 (3) | 3 (5) | 4 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 2 (3) | 1 (1)
CPK increased (Investigations) | 1 (4) | 2 (2) | 3 (7) | 5 (10)
Cardiac disorders - Other, Right Bundle Branch Block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 6 (7) | 2 (2) | 2 (3) | 4 (5)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 2 (7) | 1 (2) | 3 (4) | 4 (18)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Edema face (General disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 3 (5) | 3 (6)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 4 (7)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 5 (8) | 2 (3) | 7 (8) | 7 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (9) | 0 (0) | 1 (2) | 2 (2)
Infections and infestations - Other, Pseudomonas bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Strap epi (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Investigations - Other, PTT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (6)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (33) | 0 (0) | 16 (115) | 15 (100)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Metabolism and nutrition disorders - Other, Low C02 (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, mild neck stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Hip dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 2 (4) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mild encephalopathy with reversible splenial lesion (MERS)
Nervous system disorders - Other, eye twitching (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 12 (64) | 4 (27) | 14 (91) | 11 (82)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 11 (59) | 5 (31) | 12 (114) | 14 (203)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (1) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 3 (5) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0) | 3 (3) | 3 (4)
Respiratory, thoracic and mediastinal disorders - Other, Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (6) | 6 (7)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, erythema around insertion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, folliculitis on back (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (9) | 0 (0) | 8 (14) | 9 (19)
Weight gain (Investigations) | 6 (14) | 4 (10) | 1 (1) | 9 (19)
Weight loss (Investigations) | 4 (8) | 1 (1) | 2 (6) | 1 (2)
White blood cell decreased (Investigations) | 13 (86) | 4 (38) | 16 (121) | 13 (103)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (4) | 6 (7) | 6 (7)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 4 (5) | 1 (1) | 1 (2) | 3 (3)
Investigations - Other, Total C02 Low (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, perirectal lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 0 (0) | 6 (12) | 7 (30)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0) | 6 (15) | 7 (32)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 2 (3)
Cardiac disorders - Other, gallop (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 8 (9) | 4 (6) | 11 (17) | 7 (12)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 4 (7) | 10 (18)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 2 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Encephalitis infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, w/bilateral conjunctival hemorrhage (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 2 (2) | 3 (6) | 7 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (8) | 1 (1) | 6 (10) | 7 (15)
Fever (General disorders) | 14 (33) | 5 (19) | 14 (96) | 16 (112)
Fibrinogen decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal disorders - Other, heartburn (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, R. conjunctival hemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Genital edema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (9) | 3 (5) | 7 (21) | 9 (21)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 5 (7) | 7 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (60) | 4 (16) | 7 (33) | 7 (63)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (1) | 4 (18)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (7) | 2 (3) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 8 (16) | 1 (1) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 5 (21) | 3 (11) | 9 (50) | 7 (16)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 7 (10) | 5 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (33) | 4 (14) | 13 (62) | 16 (107)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (32) | 4 (17) | 8 (28) | 11 (30)
Hypokalemia (Metabolism and nutrition disorders) | 11 (31) | 3 (7) | 10 (63) | 13 (65)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (18) | 4 (5) | 8 (31) | 11 (29)
Hyponatremia (Metabolism and nutrition disorders) | 5 (8) | 2 (2) | 11 (28) | 15 (75)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (23) | 4 (13) | 7 (26) | 13 (110)
Hypothermia (General disorders) | 1 (5) | 1 (1) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, VRE positive (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, strap epi line inf (contaminated blood) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (5)
Investigations - Other, Low C02 (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Localized edema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Meningismus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, Bicarbonate, low (Metabolism and nutrition disorders) | 3 (11) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Mastoid inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (11) | 2 (4) | 11 (19) | 11 (25)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Nervous system disorders - Other, Still jaw (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 1 (1)
Pain (General disorders) | 5 (5) | 1 (1) | 12 (47) | 13 (48)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 5 (23) | 7 (22)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papilledema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2) | 3 (6) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — pulmonary infiltrates bilaterally
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (10)
Sinus bradycardia (Cardiac disorders) | 4 (11) | 1 (2) | 0 (0) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 7 (26) | 1 (1) | 9 (43) | 8 (23)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Dermatitis. Redness on cheeks and back.
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — redness and intermittent burning over his scrotum
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 3 (8) | 5 (10)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0) | 3 (4)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — left ventriculoperitoneal shunt
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Blood and lymphatic system disorders - Other, Thrombosis of IVC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, R sided soft tissue swelling face/neck (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, mild L foot drop when walking (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, mildly diaphoretic (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Vancomycin-resistant Enterococcus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, nasal drainage (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, oral thrush (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, C. Diff. positive (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, rhinovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, strep mitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, vesicles on R upper lip (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (3) | 3 (5)
Musculoskeletal and connective tissue disorder - Other, hypotonia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, R hand tingling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, cyclical dilatation & constriction of pupils (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, dysmetria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, gross hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, high muscle tone (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, rhinovirus/enterovirus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, splenomegaly (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, coarse breath, crackles at bilateral bases (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — petechial rash under eyes & across chest
Skin and subcutaneous tissue disorders - Other, erythema scrotum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — erythematous rash, transient
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — nasal pain, edema, erythema tip of nose (cellulitis)
Skin and subcutaneous tissue disorders - Other, erythematous rash around catheter (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, hives (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — hyperesthesia from systemic chemo infusion
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — petechiae L arm above elbow, L upper chest
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — scant erythema around bilateral eyes
Skin and subcutaneous tissue disorders - Other, slight erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, dry lips (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, skin slightly mottled (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, puffy in face and at ankles (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, upper lip swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — swelling of bilaterally submandibular regi
Infections and infestations - Other, C. Diff. (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, L. deviated gaze (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, uncontrollable blinking (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, patchy opacities in lungs (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — new lung infiltrates with this appearance in this setting may be due to infection, pulmonary edema, hemorrhage
Investigations - Other, PT prolonged (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, Lump on L. leg (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (6) | 1 (5) | 4 (6) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (5) | 0 (0) | 1 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Skin and subcutaneous tissue disorders - Other, bleeding at site of line (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT01593696/Prot_SAP_000.pdf
  • Informed Consent Form: Standard Consent (2016-05-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT01593696/ICF_001.pdf
  • Informed Consent Form: Screening Consent (2016-05-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT01593696/ICF_002.pdf